CLINICAL TRIAL: NCT04512378
Title: Facing the Unknown Together: Piloting a Group-based CBT Protocol for Intolerance of Uncertainty
Brief Title: Group CBT for Intolerance of Uncertainty
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator medical & maternity leave
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Elizabeth Hebert, Assistant Professor, University of Manitoba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2019:412
Record Dates: First submitted 2020-08-07; First posted 2020-08-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Generalized Anxiety Disorder; Intolerance of Uncertainty; Anxiety
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IU Group Treatment (Experimental): Clinical intervention arm
  Interventions: Behavioral: Behavioural Experiments for Intolerance of Uncertainty

INTERVENTIONS:
Behavioral: Behavioural Experiments for Intolerance of Uncertainty — Cognitive-behavioural treatment targeting intolerance of uncertainty using behavioural experiment technique

SUMMARY:
Generalized anxiety disorder (GAD) is a debilitating condition involving excessive and uncontrollable worry and anxiety. Difficulty tolerating the uncertainties of life, known as intolerance of uncertainty (IU), has been shown to be key in the development and maintenance of GAD symptoms. A new, streamlined cognitive-behavioural treatment that targets IU has been shown to be effective in at reducing GAD symptoms, IU, and general psychopathology when delivered one-on-one with a therapist, as shown in a recently published pilot study. The individual format of this treatment is now being evaluated in a randomized controlled trial (RCT). The overall objective of this study is to pilot test a group version of the treatment protocol to determine if a future RCT of this group treatment is both warranted and feasible. We will also conduct a preliminary investigation into the group treatment's efficacy. A total of two pilot groups (N = 12-20) will be conducted with participants recruited from two clinical hospital sites in Winnipeg, Manitoba, Canada. The group treatment protocol will be delivered over the course of 12 weekly therapy sessions. Participants will complete assessment measures at pretreatment, posttreatment, and at a 3-month follow-up point. All assessments and treatment sessions will be conducted virtually via videoconferencing platform due to ongoing COVID-19 pandemic restrictions.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of generalized anxiety disorder (GAD)
* High Intolerance of uncertainty (IU)

Exclusion Criteria:

* Comorbid psychosis, organic brain disorder, bipolar disorder, or current substance use disorder
* Receiving concurrent psychological treatments or other counselling
* Psychotropic medications must remain stable during the study period and for 3 months prior to intervention

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
MINI International Neuropsychiatric Interview | Pretreatment (prior to the intervention).
  Diagnostic status as measured by the MINI (Sheehan et al., 1994). Clinical Severity Rating adapted from the ADIS, with scores ranging from 0-8 (higher scores indicating greater GAD severity)
MINI International Neuropsychiatric Interview | Posttreatment (after completing final session of the treatment intervention)
  Diagnostic status as measured by the MINI (Sheehan et al., 1994).Clinical Severity Rating adapted from the ADIS, with scores ranging from 0-8 (higher scores indicating greater GAD severity)
MINI International Neuropsychiatric Interview | 3-month follow-up
  Diagnostic status as measured by the MINI (Sheehan et al., 1994). Clinical Severity Rating adapted from the ADIS, with scores ranging from 0-8 (higher scores indicating greater GAD severity)
Worry and Anxiety Questionnaire | Pretreatment (prior to the intervention).
  Self-reported GAD symptoms as measured by the WAQ (Dugas et al., 2001). Scores range from 0-80 with higher scores indicating higher GAD severity.
Worry and Anxiety Questionnaire | Posttreatment (after completing final session of the treatment intervention)
  Self-reported GAD symptoms as measured by the WAQ (Dugas et al., 2001). Scores range from 0-80 with higher scores indicating higher GAD severity.
Worry and Anxiety Questionnaire | 3-month follow-up
  Self-reported GAD symptoms as measured by the WAQ (Dugas et al., 2001). Scores range from 0-80 with higher scores indicating higher GAD severity.
Intolerance of Uncertainty Scale | Pretreatment (prior to the intervention).
  Self-reported difficulties tolerating uncertainty (Freeston, Rhéaume, et al., 1994). Scores range from 27-135 with greater scores indicating greater intolerance of uncertainty.
Intolerance of Uncertainty Scale | Posttreatment (after completing final session of the treatment intervention)
  Self-reported difficulties tolerating uncertainty (Freeston, Rhéaume, et al., 1994). Scores range from 27-135 with greater scores indicating greater intolerance of uncertainty.
Intolerance of Uncertainty Scale | 3-month follow-up
  Self-reported difficulties tolerating uncertainty (Freeston, Rhéaume, et al., 1994). Scores range from 27-135 with greater scores indicating greater intolerance of uncertainty.

SECONDARY OUTCOMES:
Depression Anxiety Stress Scales | Pretreatment (prior to the intervention).
  A measure of self-reported depression, anxiety, and stress symptoms (Lovibond & Lovibond, 1995). Higher scores on a subscale indicate greater severity in that symptom area (i.e., depression, anxiety, or stress, respectively).
Depression Anxiety Stress Scales | Posttreatment (after completing final session of the treatment intervention)
  A measure of self-reported depression, anxiety, and stress symptoms (Lovibond & Lovibond, 1995). Higher scores on a subscale indicate greater severity in that symptom area (i.e., depression, anxiety, or stress, respectively).
Depression Anxiety Stress Scales | 3-month follow-up
  A measure of self-reported depression, anxiety, and stress symptoms (Lovibond & Lovibond, 1995). Higher scores on a subscale indicate greater severity in that symptom area (i.e., depression, anxiety, or stress, respectively).
Penn State Worry Questionnaire | Pretreatment (prior to the intervention).
  A measure of self-reported excessive worry (Meyer, Miller, Metzger, & Borkovec, 1990). Scores range from 16-80 with higher scores indicating greater worry severity.
Penn State Worry Questionnaire | Posttreatment (after completing final session of the treatment intervention)
  A measure of self-reported excessive worry (Meyer, Miller, Metzger, & Borkovec, 1990). Scores range from 16-80 with higher scores indicating greater worry severity.
Penn State Worry Questionnaire | 3-month follow-up
  A measure of self-reported excessive worry (Meyer, Miller, Metzger, & Borkovec, 1990). Scores range from 16-80 with higher scores indicating greater worry severity.
Five Dimensional Curiosity Scale | Pretreatment (prior to the intervention).
  Self-reported tendency toward 5 dimensions of curiosity (Kashdan et al., 2018), with higher scores on each respective subscale indicating greater tendency toward a specific facet of curiousity.
Five Dimensional Curiosity Scale | Posttreatment (after completing final session of the treatment intervention)
  Self-reported tendency toward 5 dimensions of curiosity (Kashdan et al., 2018), with higher scores on each respective subscale indicating greater tendency toward a specific facet of curiousity.
Five Dimensional Curiosity Scale | 3-month follow-up
  Self-reported tendency toward 5 dimensions of curiosity (Kashdan et al., 2018), with higher scores on each respective subscale indicating greater tendency toward a specific facet of curiousity.
Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form | Pretreatment (prior to the intervention).
  Self-reported quality of life (Endicott, Nee, Harrison, & Bulmental, 1993), with scores ranging from 14-70 (higher scores indicating greater overall quality of life).
Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form | Posttreatment (after completing final session of the treatment intervention)
  Self-reported quality of life (Endicott, Nee, Harrison, & Bulmental, 1993), with scores ranging from 14-70 (higher scores indicating greater overall quality of life).
Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form | 3-month follow-up
  Self-reported quality of life (Endicott, Nee, Harrison, & Bulmental, 1993), with scores ranging from 14-70 (higher scores indicating greater overall quality of life).
Treatment Acceptability/Adherence Scale | Midtreatment
  Self-report measure of the participant's perception of the treatment's acceptability and their anticipated adherence to the intervention (Milosevic, Levy, Alcolado, & Radomsky, 2015). Scores range from 10 to 70 with greater scores indicating greater treatment acceptability and anticipated adherence.
GAD Safety Behaviours Questionnaire | Pretreatment (prior to the intervention).
  Self-reported tendency to use safety behaviours to manage anxiety (Hebert & Dugas, 2019). Scores range from 18 to 90 with higher scores indicating greater use of safety behaviours.
GAD Safety Behaviours Questionnaire | Posttreatment (after completing final session of the treatment intervention)
  Self-reported tendency to use safety behaviours to manage anxiety (Hebert & Dugas, 2019). Scores range from 18 to 90 with higher scores indicating greater use of safety behaviours.
GAD Safety Behaviours Questionnaire | 3-month follow-up
  Self-reported tendency to use safety behaviours to manage anxiety (Hebert & Dugas, 2019). Scores range from 18 to 90 with higher scores indicating greater use of safety behaviours.
IUS Past-Week | Weekly from session 1 to session 12 of treatment
  Self-report measure assessing intolerance of uncertainty in the past week (Dugas, 2008). Scores range from 27-135 with greater scores indicating greater intolerance of uncertainty in the past week.
Penn State Worry Questionnaire Past-Week | Weekly from session 1 to session 12 of treatment
  Self-report measure of the tendency to worry excessively in the past week (Stöber, J., & Bittencourt, J., 1998). Scores range from 0 to 90 with greater scores indicating greater tendency to worry excessively in the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Hebert, PhD, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Deer Lodge Centre, Winnipeg, Manitoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hebert, E. A., & Dugas, M. J. (2019). Behavioral experiments for intolerance of uncertainty: Challenging the unknown in the treatment of generalized anxiety disorder. Cognitive and Behavioral Practice, 26(2), 421-436. https://doi.org/10.1016/j.cbpra.2018.07.007
- [Background] Sheehan, D. V., Lecrubier, Y., Janvas, J., Knapp, E., Weiller, E., Sheehan, M., et al. (1994). Mini International Neuropsychiatric Interview Version 4.4 (MINI). Tampa/Paris: University of South Florida/Inserm U302-Hôpital de la Salpêtrière.
- [Background] Dugas, M. J., Freeston, M. H., Provencher, M. D., Lachance, S., Ladouceur, R., & Gosselin, P. (2001). Journal de Thérapie Comportementale et Cognitive, 11(1), 31-36.
- [Background] Meyer TJ, Miller ML, Metzger RL, Borkovec TD. Development and validation of the Penn State Worry Questionnaire. Behav Res Ther. 1990;28(6):487-95. doi: 10.1016/0005-7967(90)90135-6. PMID 2076086
- [Background] Milosevic I, Levy HC, Alcolado GM, Radomsky AS. The Treatment Acceptability/Adherence Scale: Moving Beyond the Assessment of Treatment Effectiveness. Cogn Behav Ther. 2015;44(6):456-69. doi: 10.1080/16506073.2015.1053407. Epub 2015 Jun 19. PMID 26091250
- [Background] Freeston, M. H., Rhéaume, J., Letarte, H., Dugas, M. J., & Ladouceur, R. (1994). Why do people worry? Personality and Individual Differences, 17, 791-802. https://doi.org/10.1016/0191-8869(94)90048-5
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Kashdan, T.B., Stiksma, M.C., Disabato, D., McKnight, P.E., Bekier, J., Kaji, J., & Lazarus, R. (in press). The five-dimensional curiosity scale: Capturing the bandwidth of curiosity and identifying four unique subgroups of curious people. Journal of Research in Personality
- [Background] Endicott J, Nee J, Harrison W, Blumenthal R. Quality of Life Enjoyment and Satisfaction Questionnaire: a new measure. Psychopharmacol Bull. 1993;29(2):321-6. PMID 8290681
- [Background] Stober J, Bittencourt J. Weekly assessment of worry: an adaptation of the Penn State Worry Questionnaire for monitoring changes during treatment. Behav Res Ther. 1998 Jun;36(6):645-56. doi: 10.1016/s0005-7967(98)00031-x. PMID 9648338
- [Background] Dugas, M.J. (2008). Échelle d'intolérance à l'incertitude - Dernière semaine. Montréal, Canada: Clinique des troubles anxieux, Hôpital du Sacré-Coeur de Montréal.